CLINICAL TRIAL: NCT02047214
Title: Phase 2 Dose-Escalation Study of TPI 287 in Combination With Bevacizumab in Adults With Recurrent or Progressive Glioblastoma Following a Bevacizumab-Containing Regimen
Brief Title: Safety & Efficacy Study of TPI 287 + Avastin in Adults With Glioblastoma That Progressed Following Prior Avastin Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to lack of clinical benefit in the 17 subjects enrolled in the trial to date
Sponsor: Cortice Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TPI-287-18
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma multiforme; Glioblastoma; Radiotherapy; Temozolomide; TPI 287; Taxoid; Avastin; Bevacizumab
MeSH Terms: conditions — Glioblastoma | interventions — TPI-287; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TPI 287 + bevacizumab (Experimental): All subjects will be administered TPI 287 as an IV infusion (1-hour target duration) once every 3 weeks (Days 1 and 22) and bevacizumab as a 30 to 90 minute IV infusion once every 2 weeks (Days 1, 15, and 29) of a 42-day cycle. The dose of TPI 287 will be escalated in sequential dose cohorts of 3 to 6 subjects, while the dose of bevacizumab remains constant (10 mg/kg). The planned dose escalation levels are 140, 160, 170, and 180 mg/m2; subsequent dose levels will be increased in increments of 10 mg/m2. If dose de-escalation below the starting dose level of 140 mg/m2 is required, dose levels of 130 and 120 mg/m2 will be used. Once the MTD is identified, 6 additional subjects will be enrolled at the MTD to better characterize the toxicity profile at this level. Subjects may continue on treatment unless they meet one or more of the discontinuation criteria outlined in the protocol.
  Interventions: Drug: TPI 287; Drug: Bevacizumab

INTERVENTIONS:
Drug: TPI 287 — TPI 287 is a microtubule inhibitor belonging to the taxane diterpenoid (taxoid) family, and specifically to the abeotaxane class. TPI 287 is an Investigational Drug.
  Other Names: TPI-287; NBT 287
Drug: Bevacizumab — Avastin (bevacizumab) is an FDA approved drug indicated for multiple cancers, including as a single agent for GBM for adult patients with progressive disease following prior therapy. Single agent effectiveness is based on improvement in objective response rate; no data is available demonstrating improvement in disease-related symptoms or survival with bevacizumab.
  Other Names: Avastin

SUMMARY:
The purpose of this study is to evaluate the safety, maximum tolerated dose (MTD), and efficacy of TPI 287 in combination with Avastin (bevacizumab) in subjects who have glioblastoma multiforme (GBM) that has progressed following prior radiation and temozolomide (TMZ) therapy and that has progressed following prior bevacizumab therapy.

DETAILED DESCRIPTION:
This multi-center trial is a phase 2, dose-escalation study of the safety, tolerability (MTD), and efficacy of TPI 287 in combination with bevacizumab in subjects who have GBM that has progressed following prior radiation and TMZ therapy and that has progressed following prior bevacizumab therapy.

All subjects will be administered TPI 287 as an intravenous (IV) infusion (target duration of 1 hour) once every 3 weeks (Days 1 and 22 of a 42-day cycle) and bevacizumab as a 30 to 90 minute IV infusion once every 2 weeks (Days 1, 15, and 29 of the 42-day cycle). The subsequent cycle will start 3 weeks after the last TPI 287 infusion and 2 weeks after the last bevacizumab infusion, maintaining the once every 3 week and once every 2 week schedule, respectively.

The dose of TPI 287 will be escalated in sequential dose cohorts of 3 to 6 subjects, while the dose of bevacizumab remains constant (10 mg/kg). The initial cohort of 3 subjects will be treated at a TPI 287 dose of 140 mg/m2 (dose level 0). The next dose level will be 160 mg/m2 (dose level 1). Subsequent dose levels will be increased in increments of 10 mg/m2 (i.e., dose level 2 = 170 mg/m2, dose level 3 = 180 mg/m2, etc.). If dose de-escalation below the starting dose level is required, dose levels of 130 and 120 mg/m2 will be used. Twelve (12) to 18 subjects are planned for enrollment during the dose escalation phase, depending on the number of subjects that experience dose limiting toxicities (DLTs).

Once the MTD is identified, 6 additional subjects will be enrolled at the MTD (for a total of 12) to better characterize the toxicity profile at this level.

Dose modifications and delays will be required as described in the protocol. Subjects may continue on treatment unless they meet one or more of the discontinuation criteria outlined in the protocol. Subjects who are discontinued prior to completing Cycle 1 for any reason other than toxicity will be replaced.

Adverse events (AEs) and concomitant medications will be monitored throughout the study. Subjects will be given a diary to record any AEs or concomitant medications taken between visits. Additional safety evaluations will include physical examination (including neurologic examination), Karnofsky performance status (KPS), weight (body surface area, BSA), vital signs, hematology, serum chemistry, and urinalysis.

Efficacy evaluations will include magnetic resonance imaging [MRI, including both pre and post-gadolinium T1-weighted scans and T2/fluid attenuated inversion recovery (FLAIR) images], corticosteroid usage, and neurologic status (as measured by neurologic exam and KPS).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven GBM
2. Disease progression following radiation & TMZ
3. 1st progression of GBM on bevacizumab-containing regimen or within 8 weeks of discontinuing bevacizumab. In either case, must have received a minimum of 8 weeks (4 infusions) of bevacizumab.
4. Baseline MRI must be performed after subject signs informed consent form (ICF), within 17 days of Day 1, & on steroid dosage that has been stable or decreasing for at least 5 days
5. Recent resection of recurrent or progressive tumor allowed as long as at least 4 weeks have elapsed from date of surgery & subject has recovered from surgery
6. Life expectancy >12 weeks
7. Eighteen years old or older
8. KPS equal to or greater than 70
9. Recovered from toxic effects of prior therapy to < Grade 2 toxicity per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) prior to Day 1. Minimum duration required between prior therapy & Day 1 is:

   1. At least 12 weeks from completion of radiation therapy except if there is unequivocal evidence for tumor recurrence in which case at least 4 weeks
   2. 4 weeks from prior cytotoxic therapy
   3. 4 weeks from prior experimental drug
   4. 6 weeks from nitrosoureas
   5. 3 weeks from procarbazine
   6. 1 week for non-cytotoxic agents (e.g., interferon, tamoxifen, & cis-retinoic acid)
   7. 14 days from last dose of bevacizumab
10. Adequate bone marrow function [absolute neutrophil count (ANC) > 1,500/mm3 & platelet count of > 100,000/mm3], adequate liver function [alanine aminotransferase (ALT) & aspartate aminotransferase (AST) <3 x upper limit normal (ULN), alkaline phosphatase <2 x ULN, & total bilirubin <1.5 mg/dL], & adequate renal function (BUN & creatinine <1.5 x ULN)
11. Minimum hemoglobin of 9 g/dL
12. Males & women of childbearing potential must agree to abstain from sex or use an adequate method of contraception for duration of study & for 6 months after last dose of study drug
13. Signed & dated ICF prior to Screening evaluations

Exclusion Criteria:

1. Radiographic evidence of contrast-enhancing tumor crossing midline, leptomeningeal dissemination, gliomatosis cerebri or infratentorial tumor
2. Evidence or suspicion of disease metastatic to sites remote from supratentorial brain
3. Prior treatment with anti-vascular endothelial growth factor (VEGF) drugs other than bevacizumab
4. Prior treatment with tyrosine-kinase inhibitors targeting VEGF, platelet-derived growth factor, fibroblast growth factor, tyrosine kinase with immunoglobulin-like and epidermal growth factor-like domains 2 (TIE-2), or angiopoietin (or their receptors)
5. Prior treatment with histone deacetylase inhibitors or mammalian target of rapamycin (mTOR) inhibitors
6. Prior treatment with TPI 287
7. Treatment with Enzyme-Inducing Anti-Epileptic Drugs within 2 weeks prior to Day 1
8. Treatment with drugs or herbal supplements known to be strong inhibitors/inducers of cytochrome P450 3A4 or 2C8 within 2 weeks prior to Day 1
9. Received more than one course of radiation therapy or more than a total dose of 65 Gy. May have received radiosurgery as part of initial therapy; however, dose counts against total dose limit.
10. Prior taxane, vincristine, or other microtubule inhibitor chemotherapies for treatment of GBM or other malignancy
11. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during course of study
12. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
13. Any condition, including the presence of clinically significant laboratory abnormalities, which places subject at unacceptable risk if he/she were to participate in study or confounds the ability to interpret data from study, including:

    1. Active infection including known AIDS or Hepatitis C or with a fever ≥38.5°C within 3 days prior to study enrollment
    2. Diseases or conditions that obscure toxicity or dangerously alter drug metabolism
    3. Serious intercurrent medical illness (e.g., symptomatic congestive heart failure)
14. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent subject from providing informed consent
15. Inadequately controlled hypertension (defined as systolic blood pressure >140 mmHg and/or diastolic blood pressure > 90 mmHg)
16. Prior history of hypertensive crisis or hypertensive encephalopathy
17. New York Heart Association Grade II or greater congestive heart failure
18. History of myocardial infarction or unstable angina within 6 months prior to Day 1
19. History of stroke or transient ischemic attack within 6 months prior to Day 1
20. Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
21. History of hemoptysis (≥ 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
22. Evidence of bleeding diathesis or significant coagulopathy (in absence of therapeutic anticoagulation)
23. Grade 2 or higher peripheral neuropathy per NCI CTCAE
24. History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
25. Serious, non-healing wound, active ulcer, or untreated bone fracture
26. Proteinuria at Screening. Subjects with a urine dipstick protein ≥ 2+ at Screening will undergo a 24-hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible.
27. Known hypersensitivity to any inactive ingredient of bevacizumab
28. Known hypersensitivity to any inactive ingredient of TPI 287
29. Pregnancy (positive pregnancy test) or lactation
30. Inability to comply with protocol or study procedures
31. Previously or currently enrolled in Protocol No. TPI-287-17

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety of TPI 287 + bevacizumab in adults with GBM that progressed following radiation & TMZ & prior bevacizumab as measured by AEs, physical/neurologic exam, KPS, weight, vital signs, hematology, serum chemistry, & urinalysis | Continuously over study treatment through 4 weeks after last dose of study drug
MTD of TPI 287 + bevacizumab in adults with GBM that progressed following radiation & TMZ & prior bevacizumab | Within 42 days of receiving the first dose of study drug
  The MTD will be defined as the highest dose level achieved at which no more than 1 out of 6 subjects experienced a DLT that initiated within 42 days of receiving the first dose of study drug.

SECONDARY OUTCOMES:
Efficacy of TPI 287 + bevacizumab in adults with GBM that progressed following radiation & TMZ & prior bevacizumab as measured by median progression free survival (PFS), overall response rate, & PFS rate at 4 & 6 months (PFS4 & PFS6) | Baseline & on Day 1 of each 42-day treatment cycle starting with Cycle 2, and/or as clinically indicated
  The Response Assessment in Neuro-Oncology (RANO) working group recommendations for updated response criteria for high-grade gliomas (Wen et al. 2010) will be used to determine response for this trial.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel A. Goldlust, M.D., Principal Investigator — John Theurer Cancer Center at Hackensack University Medical Center; Louis B. Nabors, III, M.D., Principal Investigator — University of Alabama at Birmingham; Sigmund Hsu, M.D., Principal Investigator — Memorial Hermann Hospital; Nimish Mohile, M.D., Principal Investigator — University of Rochester; Solmaz Sahebjam, M.D., Principal Investigator — H Lee Moffitt Cancer Center and Research Institute, Inc.; Tara L. Benkers, M.D., Principal Investigator — Swedish Neuroscience Institute; Priya Kumthekar, M.D., Principal Investigator — Northwestern University; Jian Campian, M.D., Ph.D., Principal Investigator — Washington University School of Medicine; David Schiff, M.D., Principal Investigator — University of Virginia Health System; Camilo E. Fadul, M.D., F.A.A.N., Principal Investigator — Dartmouth-Hitchcock Medical Center; Pierre Giglio, M.D., Principal Investigator — Ohio State University
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - H Lee Moffitt Cancer Center and Research Institute, Inc., Tampa, Florida
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Washington University, School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Memorial Hermann Hospital, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Swedish Neuroscience Institute, Seattle, Washington